CLINICAL TRIAL: NCT02400190
Title: The IDEA Study (Individualized Decisions for Endocrine Therapy Alone)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Rutgers Cancer Institute of New Jersey (Other); East Carolina University (Other); Stanford University (Other); Harvard University (Other); Yale University (Other); University of Pennsylvania (Other); Medical College of Wisconsin (Other); Memorial Sloan Kettering Cancer Center (Other); University of Texas Southwestern Medical Center (Other); Johns Hopkins University (Other); Loyola University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2014.111; HUM00092923 (Other: University of Michigan)
Record Dates: First submitted 2015-03-23; First posted 2015-03-26 (Estimated); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Breast Neoplasms
Keywords: radiation; lumpectomy; favorable biology; omission
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Endocrine therapy alone (Experimental): Patients receive endocrine therapy alone without radiotherapy
  Interventions: Other: endocrine therapy alone without radiotherapy

INTERVENTIONS:
Other: endocrine therapy alone without radiotherapy — Patients will not receive radiotherapy, which is the current standard for treatment for their type of breast cancer.

SUMMARY:
This study will collect rates of local/regional recurrence in select patients who do not receive radiation treatment after lumpectomy surgery. These women must be postmenopausal; have hormone receptor-positive, Her2-negative tumors; have Oncotype-DX RS less than or equal to 18; and plan to receive endocrine therapy. In this way, this study seeks to collect prospective data supporting the idea that this is a population at sufficiently low risk of local/regional recurrence that omission of adjuvant radiation might be a reasonable option.

DETAILED DESCRIPTION:
This study's primary aim is to determine rates of recurrence with the innovative approach of considering tumor biology to select patients who may avoid radiation, with restriction of eligibility to women aged 50-69 with hormone-sensitive, Her2-negative tumors with Oncotype-DX RS ≤ 18 who plan to receive endocrine therapy. In this way, this study seeks to collect prospective data supporting the idea that this is a population at low risk of LRR in whom omission of adjuvant radiation is reasonable.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal status, as defined by (a) patients age 60 or greater, or, (b) patients age 50-69 with either (a) s/p bilateral oophorectomy, or, (b) intact uterus without menses in the past 12 months, or, (c) biochemical confirmation of postmenopausal status.
* Histopathological confirmation of Stage 1 (pT1N0M0) invasive breast cancer status post breast conserving surgery
* Negative axillary nodes (isolated tumor cells with no cluster measuring >0.2mm allowed)

  * Allowable options for axillary staging include:
  * Sentinel node biopsy only
  * Sentinel node biopsy followed by axillary dissection
  * Axillary dissection only
* Margins of excision ≥2mm
* ER+, PR+, Her2 - using the current College of American Pathologists guidelines
* Oncotype-DX RS ≤ 18
* Disease must be unifocal on clinical, radiologic, and pathologic examination
* Registration within 90 days of last surgical procedure for breast cancer treatment
* Patient must willingly sign study specific informed consent prior to study entry
* Patient must be a candidate for and willing to take endocrine therapy for minimum of 5 years (aromatase inhibitor or tamoxifen). Patients who have already begun endocrine therapy after lumpectomy are eligible.
* Patient must have had breast imaging (mammogram or MRI) of the ipsilateral breast within 6 months and contralateral breast within 1 year of study entry.
* Patient must have Zubrod performance status 0-2

Exclusion Criteria:

* Evidence of multifocal or multicentric breast cancer that has not been biopsy-proven negative. Note that MRI is not required for this study, but if performed, evidence of disease beyond the site of the primary tumor in the ipsilateral breast or in the contralateral breast must be biopsy-proven not to be malignant before registration.
* Metastatic disease. Note that no specific staging studies are mandated, but any studies performed must not provide clear evidence of metastatic spread.
* Previous radiation therapy to the breast region
* Prior DCIS or invasive breast cancer
* Bilateral breast cancer
* Prior non-breast invasive malignancy other than non-melanoma skin cancer, unless there has been no evidence of disease for at least 5 years
* Known carrier of a mutation known to predispose towards breast cancer development (including BRCA-1 and BRCA-2). Note: testing for mutation status is not required for this protocol; this criterion applies only to patients who have been tested and have known carrier status.

Ages: 50 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2015-05-27 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Loco-regional Recurrence | 5 years of follow up
  All patients will be followed for their clinical outcome for at least 10 years, specifically: for development of recurrence (and site), the salvage therapy type if local disease recurs, for development of distant metastasis, and survival - both overall and breast-cancer specific.

CONTACTS AND LOCATIONS:
Overall Officials: Reshma Jagsi, M.D., Ph.D., Principal Investigator — University of Michigan
Locations (13):
- United States (13):
  - Stanford University, Stanford, California
  - Yale University, New Haven, Connecticut
  - Loyola University Medical Center, Maywood, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Harvard University, Cambridge, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Northwell Health, Lake Success, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - East Carolina University, Greenville, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Background] Mamounas EP, Tang G, Fisher B, Paik S, Shak S, Costantino JP, Watson D, Geyer CE Jr, Wickerham DL, Wolmark N. Association between the 21-gene recurrence score assay and risk of locoregional recurrence in node-negative, estrogen receptor-positive breast cancer: results from NSABP B-14 and NSABP B-20. J Clin Oncol. 2010 Apr 1;28(10):1677-83. doi: 10.1200/JCO.2009.23.7610. Epub 2010 Jan 11. PMID 20065188
- [Result] Fisher B, Anderson S, Bryant J, Margolese RG, Deutsch M, Fisher ER, Jeong JH, Wolmark N. Twenty-year follow-up of a randomized trial comparing total mastectomy, lumpectomy, and lumpectomy plus irradiation for the treatment of invasive breast cancer. N Engl J Med. 2002 Oct 17;347(16):1233-41. doi: 10.1056/NEJMoa022152. PMID 12393820
- [Derived] Jagsi R, Griffith KA, Harris EE, Wright JL, Recht A, Taghian AG, Lee L, Moran MS, Small W Jr, Johnstone C, Rahimi A, Freedman G, Muzaffar M, Haffty B, Horst K, Powell SN, Sharp J, Sabel M, Schott A, El-Tamer M. Omission of Radiotherapy After Breast-Conserving Surgery for Women With Breast Cancer With Low Clinical and Genomic Risk: 5-Year Outcomes of IDEA. J Clin Oncol. 2024 Feb 1;42(4):390-398. doi: 10.1200/JCO.23.02270. Epub 2023 Dec 7. PMID 38060195